CLINICAL TRIAL: NCT06287463
Title: A Master Protocol for the Multi-Cohort, Open-Label, Phase 1/2 Study of DCC-3084 as Monotherapy and in Combination With Other Antitumor Agents in Participants With Advanced Malignancies Driven by the MAPK Pathway
Brief Title: Study of DCC-3084 in Participants With Advanced Malignancies Driven by the Mitogen-Activated Protein Kinase (MAPK) Pathway
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCC-3084-01-001
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor; RAF Mutation; RAS Mutation; NF1 Mutation; Non-Small Cell Lung Cancer; Pancreatic Ductal Adenocarcinoma; Melanoma; BRAF Gene Mutation; CRAF Gene Mutation; Castration-Resistant Prostate Cancer (CRPC)
Keywords: Advanced malignancies
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DCC-3084 Module A Escalation Phase (ModA Part 1) (Experimental): Participants will receive DCC-3084 in ModA Part 1, Escalation Phase.
  Interventions: Drug: DCC-3084
- DCC-3084 Module A Expansion Phase (ModA Part 2) (Experimental): Participants will receive DCC-3084 in ModA Part 2, Expansion Phase.
  Interventions: Drug: DCC-3084

INTERVENTIONS:
Drug: DCC-3084 — Administered orally

SUMMARY:
This is a multicenter, Phase 1/2 clinical trial to evaluate DCC-3084 alone or in combination with other cancer therapies in participants with advanced cancers. Module A will enroll participants with advanced/metastatic solid tumors. Additional modules exploring other cancers may be added to the master protocol at a later date. Each module will be conducted in 2 parts: Part 1 (Dose Escalation) and Part 2 (Dose Expansion).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria ModA Part 1 and 2:

* Able to take oral medication
* If a female is of childbearing potential, must have a negative pregnancy test prior to enrollment and all participants agree to follow the contraception requirements
* Adequate organ function and electrolytes
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) of 0 to 1 at Screening
* Has a life expectancy of more than 6 months
* In addition to these general inclusion criteria, participants must meet all the module cohort-specific inclusion criteria

Inclusion Criteria ModA Part 1 Cohort Specific:

* Pathologically confirmed diagnosis of solid cancer and documentation of Kirsten rat sarcoma (KRAS), Harvey rat sarcoma virus (HRAS), neuroblastoma ras viral oncogene homolog (NRAS), v-raf murine sarcoma viral oncogene homolog B1 (BRAF), v-raf murine sarcoma viral oncogene homolog C1(CRAF), and/or neurofibromatosis 1 (NF1) mutation
* Have exhausted all available standard of care therapies that are known to provide benefit for the participant's condition, as judged by the Investigator

Inclusion Criteria ModA Part 2 Cohort Specific:

* Documented BRAF gene mutation
* Pathologically confirmed diagnosis with PD after at least one prior line of therapy in the advanced or metastatic setting

Exclusion Criteria:

General Exclusion Criteria ModA Part 1 and 2:

* Prior treatment with certain BRAF dimer inhibitors
* Female participant is pregnant or lactating
* Received any prior or concurrent medications or therapies known to be prohibited with DCC-3084 within 14 days
* Received any prior antitumor therapy or any investigational therapy within a specified timeframe prior to first dose of DCC-3084
* Known allergy or hypersensitivity to any component of the study drug
* Invasive malignancy within 2 years prior to the first dose of study drug other than the study indication or specific types of cancer treated with curative intent
* Have not recovered from all clinically relevant toxicities from prior therapy
* Impaired cardiac function
* History of recent thrombotic or embolic events
* Malabsorption syndrome or other illness that could affect oral absorption
* Major surgery within 28 days of the first dose of study drug
* In addition to the general exclusion criteria, participants will also be excluded based on the cohort-specific exclusion criteria

Exclusion Criteria: Module A Part 2 Cohort Specific:

• Has known co-occurring mutation of KRAS, HRAS, NRAS, NF1, epidermal growth factor receptor, Phosphoinositide-3-kinase, catalytic, alpha polypeptide (PI3KCA), or Phosphatase and TENsin homolog deleted on chromosome 10 (PTEN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLTs) (ModA Part 1) | Cycle 1 (28 days)
  DLTs reported during ModA Part 1.
Objective Response Rate (ORR) (ModA Part 2) | Start of Therapy to Progressive Disease (PD), Death Due to Any Cause, or Start of New Antitumor Therapy (Estimated up to 24 months)
  ORR is the percentage of participants with confirmed complete or partial remission based on indication specific criteria as defined in the protocol.

SECONDARY OUTCOMES:
ORR (ModA Part 1) | Start of Therapy to PD, Death Due to Any Cause, or Start of New Antitumor Therapy (Estimated up to 24 months)
  ORR is the percentage of participants with confirmed complete or partial remission based on indication specific criteria as defined in the protocol.
Progression-Free Survival (PFS) (ModA Part 1 and 2) | Start of Therapy to PD or Death Due to Any Cause (Estimated up to 24 months)
  PFS is the time from start of therapy to PD or death due to any cause.
Overall Survival (OS) (ModA Part 1 and 2) | Start of Therapy to Death Due to Any Cause (Estimated up to 36 months)
  OS is the time from start of therapy to death from any cause.
Pharmacokinetics (PK): Maximum observed plasma drug concentration (Cmax) (ModA Part 1 and 2) | Predose up to 12 hours postdose
  Cmax (ModA Part 1 and 2)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California San Francisco (UCSF) Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - SCRI HealthONE, Denver, Colorado
  - SCRI Florida Cancer Specialists, Orlando, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - SCRI Oncology Partners, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia